CLINICAL TRIAL: NCT04345198
Title: Adrenal Artery Ablation Treats Primary Aldosteronism With Resistant Hypertension (AAA-RHT)
Brief Title: Adrenal Artery Ablation for Primary Aldosteronism With Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Study Director, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA-RHT
Record Dates: First submitted 2020-04-05; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Resistant Hypertension
Keywords: resistant hypertension; aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervension (Experimental): Adrenal artery ablation is performed in PA patients with resistant hypertension.
  Interventions: Procedure: Adrenal Artery Ablation

INTERVENTIONS:
Procedure: Adrenal Artery Ablation — Intervention with adrenal artery ablation is performed in PA patients with resistant hypertension.

SUMMARY:
Primary aldosteronism(PA) is the most common endocrine cause of resistant hypertension. Surgery and medicine are the main treatment for PA by the current guidelines. However,only a small part of patients with PA meet the surgical criteria, and most of them have to take spironolactone or other antihypertensive drugs for long time. On the other side, long-term inhibition of aldosterone receptor may cause hyperkalemia, male breast hyperplasia and other adverse reactions. Moreover, hyperaldosterone is still not corrected by spironolactone, which cause extensive cerebrovascular damages even though blood pressure and blood potassium had been normalized.

With the development of adrenal vein sampling and adrenal ablation, the precise diagnosis and treatment of PA is possible. Selective adrenal artery ablation (AAA) was observed with significant decrease of blood aldosterone and blood pressure in patients with PA, which made it promissing that primary aldosteronism with resistant hypertension could be relieved by adrenal artery ablation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 30-65 years old.
* Primary aldosteronism with resistant hypertension.
* Informed consent signed and agreed to participate in this trial.

Exclusion Criteria:

* Secodary hyertension due to other causes.
* History of depression,schizophrenia or vascular dementia .
* History of cardio-cerebral vascular events such as congestive heart failure, myocardial infarction or stroke within 3 months.
* Hypohepatia (AST or AST is twice higher than the upper limit) or history of hepatitis or cirrhosis, hepatic encephalopathy.
* Renal insufficiency ( serum creatinine is 1.5 times higher than the upper limit) or history of dialysis and nephritic syndrome.
* Acute infections, tumor, severe arrhythmia, mental disorders, alcohol or medicine addiction.
* Fertile woman without contraceptives.
* Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the anti-hypertensive drugs.
* Allergic to or have contraindication to the contrast agents and alcohol.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Change of office systolic blood ptressure | 24 weeks
  Change of office systolic blood pressure compared with baseline after 24 weeks.

SECONDARY OUTCOMES:
Change of office dystolic blood pressure | 24 weeks
  Change of office dystolic blood pressure compared with baseline after 24 weeks.
Change of home systolic blood pressure | 24 weeks
  Change of home systolic blood pressure compared with baseline after 24 weeks.
Change of home diastolic blood pressure | 24 weeks
  Change of home diastolic blood pressure compared with baseline after 24 weeks.
Change of 24-h average systolic blood pressure | 24 weeks
  Change of 24-h average systolic blood pressure compared with baseline after 24 weeks.
Change of 24-h average diastolic blood pressure | 24 weeks
  Change of 24-h average diastolic blood pressure compared with baseline after 24 weeks.
Change of DDD of anti-hypertensive regimen | 24 weeks
  Change of Defined Daily Dose (DDD) of anti-hypertensive regimen compared with baseline after 24 weeks.
Change of plasma adrenal hormones | 24 weeks
  Change of plasma aldosterone and cortisol compared with baseline after 24 weeks.
Change of plasma renin levels | 24 weeks
  Change of plasma renin levels compared with baseline after 24 weeks.
Change of blood electrolytes | 24 weeks
  Change of serum potassium, natrium, and chlorine compared with baseline after 24 weeks.
Change of serum creatinine | 24 weeks
  Change of serum creatinine measured as umol/L compared with baseline after 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No